CLINICAL TRIAL: NCT06987734
Title: Neoadjuvant Sugemalimab + Chemotherapy Followed by Adjuvant Sugemalimab for Patients With Resectable Stage II-IIIA Non-small-cell Lung Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Ren Shengxiang, Prof., Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L23-385-01
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer (NSCLC)
Keywords: Neoadjuvant; NSCLC; immunotherapy; adjuvant
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perioperative immunotherapy group (Experimental): Neoadjuvant Sugemalimab + Chemotherapy Followed by adjuvant Sugemalimab
  Interventions: Drug: Neoadjuvant Sugemalimab + Chemotherapy Followed by Adjuvant Sugemalimab

INTERVENTIONS:
Drug: Neoadjuvant Sugemalimab + Chemotherapy Followed by Adjuvant Sugemalimab — Patients will receive 3-4 cycles of neoadjuvant treatment with preoperative suglizumab in combination with chemotherapy, followed by surgery. After surgery, patients will receive 1-4 cycles of platinum-containing adjuvant chemotherapy，followed by 1 year of adjuvant sugemalimab.

SUMMARY:
This is a single arm, open-label exploratory study conducted in resectable stage II-IIIA NSCLC without EGFR/ALK mutations, aiming to investigate feasibility, safety and efficacy of Sugemalimab in perioperative contexts. Twenty-five resectable stage II-IIIA patients are planned to be enrolled. The proportion of patients with squamous cell carcinoma will not less than 40%.

Combined neoadjuvant chemotherapy and immunotherapy with fixed dose of Sugemalimab 1200 mg IV Q3W + Platinum-based chemo in resectable stage II-IIIA NSCLC adult patients followed by surgery. After completion of neoadjuvant therapy (3-4 cycles) and before surgery, a tumor assessment will be done. Patients have to leave the study if there is evidence of progression in neoadjuvant therapy. Pathological response is planned to assessed after surgery. Following surgery, the patients with complete resection will receive an additional 1 year of Sugemalimab q3w. Treatment will commence as soon as clinically feasible post-surgery.

Informed consent will be obtained prior to tissue collection and genome sequencing for each participant. Primary tumour tissue will be obtained at diagnosis by biopsy such as percutaneous lung puncture biopsy, bronchoscopic biopsy or endobronchial ultrasound (EBUS) (based on clinical practice). Fresh tumour tissue was collected after surgical resection. Tissues collected were subjected to medically necessary pathology for diagnosis. Specimens were processed for multiplex immunofluorescence, single-cell sequencing and spatial transcriptomics, bulk RNAseq and WES to explore the changes in the immune microenvironment before and after suglizumab administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients have voluntarily to join the study and give written informed consent for the study.
3. Histologically documented, stage II-IIIA Non-Small Cell Lung Cancer (according to version 9th of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology) and previously untreated.
4. Tumor should be considered resectable before study entry by a multidisciplinary team.
5. ECOG Performance Status of 0 or 1
6. At least 1 unidimensional measurable lesion meeting Response Evaluation Criteria in Solid Tumours (RECIST) criteria.
7. Able to comply with study and follow-up procedures
8. Major organ function For regular test results（no blood transfusion within 14 days）：

   1. Hemoglobin（HB）≥90g/L；
   2. Absolute neutrophils count（ANC）≥1.5×109/L；
   3. Blood platelets（PLT）≥100×109/L

   Biochemical tests results defined as follows:
   1. Total bilirubin（TBIL）≤1.5 times the upper limit of normal (ULN) ；
   2. Alanine aminotransferase (ALT) and aspartate aminotransgerase AST≤2.5*ULN,
   3. Creatinine（Cr）≤1.5*ULN or Creatinine Clearance rate (CCr)≥60 ml/min; Coagulation test: INR/APTT within normal limits Doppler ultrasound assessment：left ventricular ejection fraction (LVEF) ≥the lower limit of normal value (50%).
9. The patients need to have a forced expiratory volume (FEV1) ≥ 1.2 liters
10. Subjects must provide fresh tissues or formalin-fixed tumor tissue samples at or the diagnosis NSCLC for mIF.

Exclusion Criteria:

* 1) All patients carrying activating mutations in the TK domain of EGFR or any variety of alterations in the ALK gene.

  2) Small cell lung cancer (including patients with mixed small cell lung cancer and non-small cell lung cancer).

  3) Any anti-tumor treatment within the past 5 years, including chemotherapy, radiotherapy, target therapy or other immunotherapy 4) Severe acute or chronic infections, including: hepatits B, hepatits C, HIV etc 5) Patients with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement or unexpected conditions of recurrence in the absence of an external trigger are allowed to be included.

  6) Histologically confirmed adenosquamous carcinoma 7) Any prior treatment of antibody/drug that targets at T-cell coregulatory proteins 8) Subjects have interstitial lung disease (ILD), or a history of ILD that required corticosteroid treatment.

  9) Women in pregnancy or lactation. 10) Patients who are allergic to any of the agent or any ingredient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response | Assessment of postoperative pathology within 6 weeks of neoadjuvant therapy
  Major Pathological Response (≤10% residual viable tumor cells in the primary tumor and sampled lymph nodes)

SECONDARY OUTCOMES:
Pathological Complete Response | Assessment of postoperative pathology within 6 weeks of neoadjuvant therapy
  0% residual viable tumor cells in the primary tumor and sampled lymph nodes
Event-free survival rate | 6 /12 /18 months
  Event-free survival rate at 6 /12 /18 months

OTHER OUTCOMES:
Analysis of the tumour immune microenvironment | Perioperative
  Specimens were processed for multiplex immunofluorescence, single-cell sequencing and spatial transcriptomics, bulk RNAseq and WES to explore the changes in the immune microenvironment before and after suglizumab administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China, Shanghai, Shanghai Municipality, China